CLINICAL TRIAL: NCT03978780
Title: Quality of Recovery Scores Following Erector Spinae Block vs. Sham Block in Ambulatory Breast Cancer Surgery: A Randomised Controlled Trial
Brief Title: Erector Spinae Block vs. Placebo Block Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0048-B
Record Dates: First submitted 2019-03-25; First posted 2019-06-07 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Nerve Block; Regional Anesthesia; Neuromuscular Blockade
Keywords: Spinae fascial plane block; Breast surgery; interfascial plane block; erector spinae block
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be a prospective, double-blinded, randomised controlled trial conducted at Women's College Hospital. The study will enroll patients undergoing unilateral breast cancer surgery involving sentinel lymph node biopsy, axillary lymph node dissection and total axillary lymph node clearance. After obtaining written informed consent from eligible patients, study participants will be randomly assigned to one of two groups, the Erector spinae block group and the Control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinded for patient, assessor, anesthesiologist in the operating room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Patients randomised to the Control group will then receive a sham subcutaneous injection of 0.5ml normal saline injected at the same site as the ESP block (see above) under ultrasound guidance to stimulate a real block procedure.
  Interventions: Procedure: Placebo Block
- Erector spinae plane (ESP) block group (Experimental): Local anaesthetic infiltration utilising 1% lidocaine will occur, and an 80mm 22G block needle will be inserted using an in-plane cranial to caudad approach, the needle will be advanced to target the interfascial plane deep to the erector spinae muscle at the T2 transverse process. Once the needle tip is in the correct position, 20 ml of the local anaesthetic (ropivacaine 0.5% with 1:400,000 epinephrine) will be administered slowly in 5 ml aliquots under frequent aspiration and correct spread in the interfascial plane will be observed.
  Interventions: Procedure: Erector spinae plane block

INTERVENTIONS:
Procedure: Erector spinae plane block — 80mm 22G block needle will be inserted using an in-plane cranial to caudad approach, the needle will be advanced to target the interfascial plane deep to the erector spinae muscle at the T2 transverse process. Once the needle tip is in the correct position, 20 ml of the local anaesthetic (ropivacaine 0.5% with 1:400,000 epinephrine) will be administered slowly in 5 ml aliquots under frequent aspiration and correct spread in the interfascial plane will be observed.
  Arms: Erector spinae plane (ESP) block group
Procedure: Placebo Block — Patients randomised to the Control group will then receive a sham subcutaneous injection of 0.5ml normal saline injected at the same site as the ESP block under ultrasound guidance to stimulate a real block procedure.
  Arms: Control Group

SUMMARY:
Regional anaesthesia combined with general anaesthesia has become common in the perioperative management of breast cancer surgery patients. Regional techniques have been recognised to provide excellent post-operative analgesia. It enhances multi-modal analgesia regimes while being opioid sparing, reducing incidence of post-operative nausea and vomiting and allowing earlier mobilisation/discharge and improving treatment success. Therefore identifying the correct regional anaesthetic technique for this group of patients is important in providing optimum peri-operative care.

DETAILED DESCRIPTION:
The ultrasound-guided erector spinae plane (ESP) block has been recently described for the successful management of thoracic neuropathic pain. The erector spinae muscle is formed by the spinalis, longissimus thoracis, and iliocostalis muscles that run vertically in the back. The ESP block is performed by depositing the local anaesthetic in the fascial plane, deep to the erector spinae muscle, at the tip of the transverse process of the vertebra. Indirect access to the paravertebral space is gained providing analgesia without the risk of needle injury to structures in close proximity. Cadaveric studies have shown both ventral and dorsal rami of thoracic spinal nerves are affected when local anaesthetic is injected deep to the erector spinae muscle. The erector spinae muscle extends along the thoracolumbar spine allowing extensive cranio-caudal spread. The ventral ramus (intercostal nerve) is divided into the anterior and lateral branches. Its terminal branches provide the sensory innervation of the entire anterolateral wall. The dorsal ramus is divided into 2 terminal branches and it gives the sensory innervation to the posterior wall. Anterior spread of the local anaesthetic to the paravertebral space through the costotransverse foramina and the intertransverse complex provides both visceral and somatic analgesia.

While recent evidence supports statistically significant reductions in pain and opioid consumption among patients who receive an ESP block compared to systemic analgesia alone, the clinical significance of these differences are questionable the effect of ESP block on the patients' quality of recovery following ambulatory breast cancer surgery remains unclear.

Therefore, our objective is to determine whether or not the addition of an ESP block provides both superior analgesia and quality of recovery in patients undergoing ambulatory breast cancer surgery compared to systemic analgesia alone. We hypothesis that patients who received a preoperative ESP block will afford superior postoperative analgesia and improve the quality of recovery over the first 24 hours following surgery compared to those who receive a sham block for their ambulatory breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA classification: I-III
* BMI < 35 kg/m2
* Day surgery procedure

Exclusion Criteria:

* Prior ipsilateral breast surgery, excluding lumpectomy
* Pre-existing neurological deficit or peripheral neuropathy involving the ipsilateral chest
* Severe, poorly controlled cardiac conditions, significant arrhythmias, severe valvular heart diseases
* Severe, poorly controlled respiratory conditions (severe COPD, severe interstitial lung disease, severe / poorly controlled asthma)
* Contraindication to regional anaesthesia (e.g. bleeding diathesis, coagulopathy, sepsis, infection at the site of potential needle puncture on the posterior chest)
* Patient refusal
* Chronic pain disorder
* Chronic opioid use (≥30 mg oxycodone / day)
* Contraindication (or allergy) to a component of multi-modal analgesia protocol
* Allergy to amide local anaesthetics used in nerve blocks
* Contraindications to any of the components of the standardized general anaesthesia
* Significant psychiatric disorder that would preclude objective study assessment
* Pregnancy/ women with nursing infants
* Unable to provide informed consent
* Unable to speak and read English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Acute postoperative pain at rest | 24 hours postoperatively
  Following breast surgery, measured as an area under the curve (AUC) of rest pain scores VAS scale where 0 corresponds to no pain, and 10 corresponds to worst pain imaginable
Quality of postoperative recovery (QoR 15) | 24 hours post-surgery
  Quality of recovery at 24 hours: questionnaire (0-10, where 0 = none of the time [poor] and 10 = all of the time [excellent])

SECONDARY OUTCOMES:
Postoperative pain scores | 0, 6, 12, 18, 24 and 48 hours post-operatively
  VAS scale where 0 corresponds to no pain, and 10 corresponds to worst pain imaginable
Intraoperative opioid consumption | During the procedure
  Cumulative oral morphine equivalent after surgery
Postoperative opioid consumption | 12,24,48 hours, 7 days postoperative
  Cumulative oral morphine equivalent after surgery
Duration of phase I (PACU) and phase II (surgical day care, SDC) stay | From end of surgical procedure to 24 hours after surgery
  How fast is the recovery is-expressed in minutes
Opioid-related side effects | End of surgical procedure to 48 hours after surgery
  Risk of opioid-related side effects(nausea, vomiting, pruritis)
Persistent post surgical pain DN4 screening tool | 3 months post operatively
  Satisfaction with pain management. Is prescribed pain medication enough?
Block-related complications | End of surgical procedure to 48 hours after surgery
  bruising at injection site, numbness over lateral chest, weakness of shoulder or arm, pain/swelling at injection site

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brull, MD,FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada